CLINICAL TRIAL: NCT02975141
Title: Gemcitabine and Nab-Paclitaxel Combined With the Oral Irreversible ErbB Family Blocker Afatinib in Patients With Metastatic Pancreatic Cancer: A Phase Ib Trial
Brief Title: Afatinib and Gemcitabine/Nab-paclitaxel in Metastatic Pancreatic Cancer
Acronym: AFFECT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PD Dr. med. Volker Heinemann (Other)
Collaborators: Technical University of Munich (Other); University of Cologne (Other)
Responsible Party: Sponsor-Investigator, PD Dr. med. Volker Heinemann, Professor of Medicine, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015-004065-86
Record Dates: First submitted 2016-09-21; First posted 2016-11-29 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Palliative Chemotherapy; Afatinib; Gemcitabine; nab-paclitaxel; pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Afatinib; Gemcitabine; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Afatinib 40Mg Tab, Gemzar, Abraxane +1 (Experimental): Dose Level +1 Afatinib 40 mg Nab-paclitaxel 125 mg/m2 BSA Gemcitabine 1000 mg/m2 BSA
  Interventions: Drug: Afatinib 40Mg Tab; Drug: Gemzar; Drug: Abraxane
- Afatinib 30Mg Tab, Gemzar, Abraxane 0 (Experimental): Dose Level 0 Afatinib 30 mg Nab-paclitaxel 125 mg/m2 BSA Gemcitabine 1000 mg/m2 BSA
  Interventions: Drug: Afatinib 30Mg Tab; Drug: Gemzar; Drug: Abraxane
- Afatinib 30Mg Tab, Gemzar, Abraxane -1 (Experimental): Dose Level -1 Afatinib 30 mg Nab-paclitaxel 100 mg/m2 BSA Gemcitabine 800 mg/m2 BSA
  Interventions: Drug: Afatinib 30Mg Tab; Drug: Gemzar; Drug: Abraxane
- Afatinib 30Mg Tab, Gemzar, Abraxane -2 (Experimental): Dose Level -2 Afatinib 30 mg Nab-paclitaxel 75 mg/m2 BSA Gemcitabine 600 mg/m2 BSA
  Interventions: Drug: Afatinib 30Mg Tab; Drug: Gemzar; Drug: Abraxane

INTERVENTIONS:
Drug: Afatinib 30Mg Tab — Study Drug
  Other Names: Giotrif
  Arms: Afatinib 30Mg Tab, Gemzar, Abraxane -1; Afatinib 30Mg Tab, Gemzar, Abraxane -2; Afatinib 30Mg Tab, Gemzar, Abraxane 0
Drug: Afatinib 40Mg Tab — Study Drug
  Other Names: Giotrif
  Arms: Afatinib 40Mg Tab, Gemzar, Abraxane +1
Drug: Gemzar — Chemotherapy Backbone
  Other Names: Gemcitabine
Drug: Abraxane — Chemotherapy Backbone
  Other Names: nab-Paclitaxel

SUMMARY:
This study sets out to determine the maximum tolerated dose (MTD) of afatinib in combination with gemcitabine/nab-paclitaxel in patients with metastatic pancreatic ductal adenocarcinoma. The identified MTD will serve as recommended phase II dose (RP2D).

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC) remains an almost uniformly lethal disease. Although there has been significant progress in understanding of the underlying molecular biology of pancreatic cancer, this progress has not translated into substantially better treatments. Alarmingly, the number of pancreatic cancer cases is constantly rising and pancreatic cancer will be the second most frequent cause of cancer related death by 2030.

Accordingly, novel therapeutic strategies for patients with pancreatic cancer are desperately needed.

Recently, the combination of gemcitabine and nab-paclitaxel proofed to be superior when compared to single agent gemcitabine (overall survival [OS] 8.7 months in the nab-paclitaxel/gemcitabine group versus 6.6 months in the gemcitabine group; hazard ratio for death, 0.72; 95% confidence interval [CI], 0.62 to 0.83; P<0.001). Consequently, this combination therapy is now regarded as a novel treatment option for patient with metastatic pancreatic cancer and should therefore serve as a backbone for future clinical studies.

Preclinical studies suggest a significant role for ErbB signaling in the pathogenesis of pancreatic cancer. Accordingly, targeting the family of ErbB receptor tyrosine kinases seems to be a viable option to improve the outcome of patients with pancreatic cancer. Addition of the selective reversible EGFR tyrosine kinase inhibitor erlotinib to gemcitabine significantly improved progression-free survival and overall survival in metastatic pancreatic cancer patients. However, the effect on median survival time in absolute values between the two arms (erlotinib and gemcitabine versus gemcitabine alone) accounted for less than a half month.

Afatinib is a selective, potent and irreversible ErbB family blocker. Unlike erlotinib, afatinib covalently binds to and irreversibly blocks signalling from all homo- and heterodimers formed by the ErbB family members EGFR (ErbB1), HER2 (ErbB2), ErbB3 and ErbB4. Afatinib is applied orally once daily. Preclinical studies suggest that application of afatinib should result in greater efficacy against tumor growth than application of erlotinib.

Afatinib as monotherapy has a marketing authorization for the treatment of locally advanced or metastatic non-small cell lung cancer (NSCLC) with activating EGFR mutation/mutations for daily doses up to 50 mg once daily. In a Phase I trial for safety and tolerability of afatinib in combination with gemcitabine in patients with advanced solid tumors the maximum tolerated dose (MTD) was 40 mg afatinib (given continuously once daily) plus 1000 mg/m2 gemcitabine on D1 and D8 of a 21-day cycle, with no dose-limiting toxicity in the respective cohort. Accordingly, in another current Phase II trial of the sponsor for treatment of metastatic pancreatic cancer the dose of 40 mg continuously orally once daily given afatinib in combination with 1000 mg/m2 gemcitabine given on Day1, Day 8, and Day 15 of a 28-day cycle against monotherapy with gemcitabine 1000 mg/m2 is used.

The investigators hypothesize that addition of afatinib to gemcitabine/nab-paclitaxel might result in better anti-tumor activity.

Accordingly, the aim of this trial is to establish the MTD for afatinib in combination with gemcitabine/nab-paclitaxel in order to proceed into Phase II trials.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥ 18 years of age and ≤ 75 years
2. Histologically (not cytologically) confirmed diagnosis of metastatic pancreatic ductal adenocarcinoma (PDAC) [Stage IV according to UICC TNM edition 7 of 2009: each T, each N, M1]
3. No option for surgical resection or radiation in curative intent
4. At least one unidimensionally measurable tumor lesion (according to RECIST 1.1)
5. ECOG performance status 0 - 1
6. Life expectancy at least 3 months
7. Adequate hepatic, renal and bone marrow function, defined as:

   * Absolute neutrophil count (ANC) ≥ 1.5x109/L
   * Haemoglobin ≥ 9 g/dL 9
   * Thrombocytes ≥100x10/L
   * Total bilirubin ≤ 1.5xULN.

     * Patients with a biliary stent may be included provided that bilirubin level after stent insertion decreased to ≤ 1.5 x ULN and there is no cholangitis.
   * AST/GOT and/or ALT/GPT ≤ 2.5 x ULN or in case of liver metastasis ≤ 5 x ULN)
   * Serum creatinine within normal limits or creatinine clearance ≥60 mL/min/1.73 m2 as calculated by CKD- EPI formula for patients with serum creatinine levels above or below the institutional normal value.
8. Acceptable coagulation studies defined as prothrombin time (or INR) and PTT ≤ 1.5 x ULN
9. Stable/decreasing pain symptoms under pain medication or no pain within the last 2 weeks before first application of study medication (as reported and assessed by the patient).
10. Females of childbearing potential (FCBP) must have a negative highly sensitive serum pregnancy test within 7 days of the first application of study treatment and they must agree to undergo a further pregnancy tests at monthly intervals and at the end of treatment visit and FCBP must either agree to use and be able to take highly effective contraceptive birth control methods (Pearl Index < 1) or agree to practice complete abstinence from heterosexual intercourse during the course of the study and for at least 1 month after last application of study treatment. A female subject following menarche is considered to be of childbearing potential unless she is naturally amenorrhoeic for ≥ 1 year without an alternative medical reason, or unless she is permanently sterile.
11. Males must agree to use condoms during the course of the trial and for at least 6 months after last administration of study drugs or practice complete abstinence from heterosexual intercourse.
12. Signed and dated informed consent before the start of any specific protocol procedures
13. Patient's legal capacity to consent to study participation

Exclusion Criteria:

1. Locally advanced PDAC without metastasis
2. Evidence of ascites
3. Known metastatic disease to the brain. Brain imaging is required in symptomatic patients to rule out brain metastases, but is not required in asymptomatic patients.
4. Previous palliative chemotherapy or other palliative systemic tumor therapy for metastatic disease of PDAC
5. Previous gemcitabine treatment with exception of gemcitabine treatment applied as monotherapy in the adjuvant setting (after potential curative R0 or R1 resection) and if the adjuvant single-agent gemcitabine chemotherapy was terminated at least 6 months before study entry
6. Previous radiotherapy of PDAC
7. Previous ErbB family directed therapy for PDAC (e. g. erlotinib, cetuximab, trastuzumab, lapatinib)
8. Any major surgery within the last 4 weeks before study entry
9. Clinical significant decrease in performance status within 2 weeks of intended first application of study medication (by medical history)
10. Severe tumor-related cachexia and/or known weight loss >15% within one month before study enrollment
11. Pre-existing polyneuropathy ≥ grade 2 according to CTCAE version 4.03
12. LDH >2.5xULN
13. Significant (≥ 20%) decrease in serum albumin levels within 2 weeks of intended first application of study medication (by medical history)
14. Gastrointestinal disorders that might interfere with the absorption of the study drug and gastrointestinal disorders with diarrhoea as a major symptom (e.g. Crohn's disease, malabsorption), and chronic diarrhoea of any aetiology CTCAE version 4.03 grade ≥ 2
15. Medical history of interstitial lung disease (ILD) or pulmonary fibrosis or severe COPD
16. Liver cirrhosis Child-Pugh other than class A
17. Known coagulopathy or bleeding disorder
18. History of connective tissue disorders (e.g. lupus, scleroderma,arteritis nods)
19. Any other severe concomitant disease or disorder, which could influence patient's ability to participate in the study and his/her safety during the study or interfere with interpretation of study results e.g. active infection, uncontrolled hypertension, clinically significant cardiovascular disease e.g. cerebral vascular accident (≤ 6 months before study start), myocardial infarction (≤ 6 months before study start), unstable angina, heart failure ≥ NYHA functional classification system grade 2, severe cardiac arrhythmia requiring medication, metabolic dysfunction, severe renal disorder.
20. Any other malignancies than PDAC within the last 5 years before study start, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer
21. Hypersensitivity to afatinib, nab-paclitaxel, or gemcitabine or to any of the excipients or to compounds with similar chemical or biologic composition
22. Continuing abuse of alcohol,drugs,or medical drugs
23. Pregnant or breast-feeding females or FCBPs unable to either perform highly effective contraceptive measures or practice complete abstinence from heterosexual intercourse
24. Current or recent (within 4 weeks prior to first application of study treatment) treatment with an investigational drug or participation in an investigational clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-09; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
MTD of afatinib in combination with gemcitabine/nab-paclitaxel | 28 days after the first dose of chemotherapy
  Completion of the first cycle of chemotherapy

SECONDARY OUTCOMES:
RECIST measurements of target lesions (in cm/inches) | 18 months
  Objective Response Rate
Progression free survival (in months) | 18 months
  PFS
Overall survival (in months) | 18 months
  OS
Incidence of Treatment-Emergent Adverse Events | 18 months
  Type, incidence, and severity of adverse events according to NCI CTCAE version 4.03. Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Volker Heinemann, Professor, Principal Investigator — University of Munich - Klinikum Großhadern
Locations (1):
- Ludwig-Maximilians - University of Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: No